CLINICAL TRIAL: NCT01577446
Title: Narrow QRS Ischemic Patients Treated With Cardiac Resynchronization Therapy
Brief Title: Narrow QRS Ischemic Patients Treated With Cardiac Resynchronization Therapy (NARROW CRT)
Acronym: NARROW-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Santa Maria di Loreto Mare (Other)
Responsible Party: Principal Investigator, Carmine Muto, Electrophysiology and Pacing Unit Director, Ospedale Santa Maria di Loreto Mare
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LM-002
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Heart Failure, Systolic
Keywords: CRT; heart failure; narrow QRS; dyssynchrony
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- CRT (Experimental): The CRT group undergoes implantation of a CRT defibrillator
  Interventions: Procedure: cardiac resynchronization therapy
- no-CRT (No Intervention): The no-CRT group receives a dual-chamber defibrillator

INTERVENTIONS:
Procedure: cardiac resynchronization therapy — Implantation of a CRT defibrillator with a standard right atrial, right ventricular defibrillator and left ventricular leads
  Arms: CRT

SUMMARY:
Current recommendations require a QRS duration of ≥120ms as a condition for prescribing cardiac resynchronization therapy (CRT). This study was designed to test the hypothesis that patients with heart failure of ischemic origin, current indications for defibrillator implantation and QRS <120ms may benefit from CRT in the presence of marked mechanical dyssynchrony.

ELIGIBILITY:
Inclusion Criteria:

* NHYA class II-III heart failure
* ischemic cardiomyopathy
* ejection fraction of 35% or less
* QRS interval of 120ms or less
* evidence of mechanical dyssynchrony as measured on echocardiography

Exclusion Criteria:

* conventional indication for cardiac pacing
* persistent atrial fibrillation
* life expectancy lower than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
heart failure clinical composite score | 12 months
  Patients are classified according to a score, which assigns subjects to one of three response groups - improved, worsened, or unchanged. Patients are judged to be worsened if they died or were hospitalized because of worsening heart failure (at any time during the 12 months), or demonstrated worsening in NYHA functional class at their 12-month visit. Patients are judged to be improved if they had not worsened and had demonstrated improvement in NYHA functional class at 12 months. Patients who are not worsened or improved are classified as unchanged.

SECONDARY OUTCOMES:
time to the first heart failure hospitalization or death | up to 30 months
  Kaplan-Meier analysis is used to analyze time to death or first heart failure hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Muto, MD, Study Chair — Ospedale Santa Maria di Loreto Mare
Locations (1):
- Ospedale Santa Maria di Loreto Mare, Naples, Italy

REFERENCES:
- [Derived] Muto C, Solimene F, Gallo P, Nastasi M, La Rosa C, Calvanese R, Iengo R, Canciello M, Sangiuolo R, Diemberger I, Ciardiello C, Tuccillo B. A randomized study of cardiac resynchronization therapy defibrillator versus dual-chamber implantable cardioverter-defibrillator in ischemic cardiomyopathy with narrow QRS: the NARROW-CRT study. Circ Arrhythm Electrophysiol. 2013 Jun;6(3):538-45. doi: 10.1161/CIRCEP.113.000135. Epub 2013 Apr 16. PMID 23592833